CLINICAL TRIAL: NCT05357781
Title: Immunoglobulin Deficiency a Treatable Cause of Fatigue in Patients With Multiple Sclerosis (MS)? - A Prospective Observational Fatigue Trial
Brief Title: Immunoglobulin Deficiency a Treatable Cause of Fatigue in Patients With Multiple Sclerosis (MS)?
Acronym: FatIgG
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-02372
Record Dates: First submitted 2022-04-19; First posted 2022-05-03 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Hypogammaglobulinemia; Multiple Sclerosis; Fatigue
Keywords: Fatigue; Hypogammaglobulinemia
MeSH Terms: conditions — Agammaglobulinemia; Multiple Sclerosis; Fatigue | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MS patients with IgG deficiency (serum IgG-concentration <7g/L).: MS patients with IgG deficiency (serum IgG-concentration <7g/L).
  Interventions: Diagnostic Test: Laboratory test
- MS patients with normal IgG serum concentration (serum IgG-concentration ≥7g/L).: MS patients with normal IgG serum concentration (serum IgG-concentration ≥7g/L).
  Interventions: Diagnostic Test: Laboratory test

INTERVENTIONS:
Diagnostic Test: Laboratory test — Frequency of fatigue (defined as Fatigue Scala for Motor and Cognitive Function (FSMC) total ≥ 43 points) in MS patients with IgG-deficiency
  Other Names: Fatigue Score

SUMMARY:
The investigators hypothesize that hypogammaglobulinemia (defined as IgG serum concentration <7.0g/L) is a treatable cause of fatigue in people with MS:

The primary objective is to prove the link between hypogammaglobulinemia and fatigue in patients with multiple sclerosis.

The secondary objective is to show that fatigue is mediated via frequent infections in people with MS and hypogammaglobulinemia.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is the most common cause of mental and physical disability in young adults affecting approximately 10'000-15'000 persons in Switzerland (incidence 16/100000; prevalence 190/100000). MS-fatigue affects at least 75% of the MS-patients (affected persons in Switzerland 7500-11250). MS-related fatigue has socioeconomic consequences leading to increased sick leaves and a higher probability of unemployment. Effective treatment strategies for MS-fatigue are missing, despite the appearance of more effective immunotherapies to treat autoimmune neuroinflammation and to control MS disease activity. The reason for the lack of therapeutic options is the unclear pathophysiological mechanism of fatigue with many non-MS associated influencing factors like thyroid dysfunction and anaemia.

Fatigue is also present in other inflammatory diseases, cancers and immunodeficiency syndromes. Regarding the latter patients with primary immunodeficiencies (PIDs) and common variable immunodeficiency (CVID) suffer from fatigue in 30 - 76%, which is more common than in the normal population. Studies investigating immunoglobulin replacement therapy in patients with CVID demonstrated a correlation between the frequency of infusions / s.c. applications and wear-off effect/fatigue.

Immunoglobulin deficiency seems to be much more common in people with autoimmune diseases. In MS reduced serum immunglobulin G (IgG) concentrations regardless of immunotherapy affect between 8 - 26% of the patients. Nonetheless consequences of IgG hypogammaglobulinemia in MS are partly unknown. However, based on the findings in patients with CVID, fatigue might be one of them. To close this knowledge gap prospective observational studies are needed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis following McDonald 2017-Criteria
* Age 18-65 years
* Stable MS disease at inclusion (definition: no clinical relapse, no MRI activity, stable disability within the last 12 months)
* Unchanged immunotherapy within the last 12 months
* Expanded Disability Status Scale (EDSS) level <4 points indicating fully ambulatory patients.
* Capability of written informed consent

Exclusion Criteria:

* Severe depression (definition: Beck Depression Index-II (BDI-II) ≥29 points) or other established psychiatric diagnosis
* Immunodeficiency other than hypogammaglobulinemia
* Immunglobulin replacement therapy or indication for immunoglobulin replacement therapy
* Severe Sleepiness (definition: Epworth-Sleepiness-Scale (ESS) >16 points)
* Fatigue aggravating factors such: liver/renal/thyroid dysfunction, substance abuse, medication (tranquilizers /antiepileptics/psychopharmaceuticals), chronic infectious disease (like hepatitis/HIV).
* Other neurodegenerative/autoimmune disease.
* Patients not able to give written consent
* Vulnerable patients such as children, pregnant women and prisoners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple Sclerosis Patients
Sampling Method: Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with fatigue and hypogammaglobulinemia | 1.5 years
  The primary endpoint will be measured as frequency (%) of fatigue (defined as Fatigue Scala for Motor and Cognitive Function (FSMC) total ≥ 43 points) in MS patients with IgG-deficiency (IgG serum concentration <7.0 g/L) compared to those with normal IgG-serum concentration (≥ 7.0 g/L).
  The FSMC is an assessment of MS-related cognitive and motor fatigue. A Likert-type 5-point scale (ranging from 'does not apply at all' to 'applies completely') produces a score between 1 and 5 for each scored question. Thus minimum value is 20 (no fatigue at all) and maximum value is 100 (severest grade of fatigue) FSMC Sum Score: ≥ 43 points mild fatigue, ≥ 53 points moderate fatigue, ≥ 63 severe fatigue
Number of patients with fatigue without hypogammaglobulinemia | 1.5 years
  The primary endpoint will be measured as frequency (%) of fatigue (defined as Fatigue Scala for Motor and Cognitive Function (FSMC) total ≥ 43 points) in MS patients with IgG-deficiency (IgG serum concentration <7.0 g/L) compared to those with normal IgG-serum concentration (≥ 7.0 g/L).
  The FSMC is an assessment of MS-related cognitive and motor fatigue. A Likert-type 5-point scale (ranging from 'does not apply at all' to 'applies completely') produces a score between 1 and 5 for each scored question. Thus minimum value is 20 (no fatigue at all) and maximum value is 100 (severest grade of fatigue) FSMC Sum Score: ≥ 43 points mild fatigue, ≥ 53 points moderate fatigue, ≥ 63 severe fatigue

SECONDARY OUTCOMES:
Fatigue and infections | 1.5 years
  As secondary endpoint the frequency of infections (infection/months) in MS patients will be measured and compared between those with (IgG serum concentration <7.0 g/L) and without hypogammaglobulinemia (IgG serum concentration ≥ 7.0 g/L). Furthermore, the mediation of fatigue by "frequency of infections*" will be detailed in the cohort of MS patients with hypogammaglobulinemia.
  *A telephone interview with 6 questions about the frequency of infections will take place once a month.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Diem, MD, Principal Investigator — Inselspital University Hospital of Bern
Locations (1):
- University Hospital of Bern Inselspital, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No